CLINICAL TRIAL: NCT03854266
Title: Low Dose Catheter Directed Thrombolysis for Acute Intermediary-high Risk Pulmonary Embolism
Brief Title: Low Dose Catheter Directed Thrombolysis for Acute Pulmonary Embolism
Acronym: BETULA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190580-0001
Record Dates: First submitted 2019-02-05; First posted 2019-02-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Catheter directed thrombolysis (Experimental): Low dose alteplase (4/8 milligram) will be infused over 2 hours locally in the pulmonary arteries at the site of the thrombus through an infusion catheter with sideholes (Unifuse, AngioDynamics, US)
  Interventions: Drug: Low dose alteplase; Device: Infusion catheter
- Unfractionated heparin (Active Comparator): Initial dose of unfractionated heparin is 80 international units per kilo (IU/kg) bolus followed by 18 IU/kg as continuous infusion with dose adjustment every 6 hours and once daily when activated partial thromboplastin time is 1.5-2.3 times control value.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Low dose alteplase — Low dose alteplase is 4 milligram per pulmonary artery (maximum dose 8 milligram) infused in the pulmonary arteries over 2 hours
  Other Names: alteplase
  Arms: Catheter directed thrombolysis
Drug: Unfractionated heparin — Unfractioned heparin is administered in a peripheral vein with an initial dose of 80 international units per kilo (IU/kg) bolus followed by 18 IU/kg as continuous infusion with dose adjustment every 6 hours and once daily when activated partial thromboplastin time (APPT) is 1.5-2.3 times control value.
  Other Names: heparin
  Arms: Unfractionated heparin
Device: Infusion catheter — A sidehole catheter (Unifuse, AngioDynamics, US) catheter will be advanced to the pulmonary arteries to facilitate the catheter directed thrombolysis
  Other Names: Unifuse
  Arms: Catheter directed thrombolysis

SUMMARY:
BETULA trial will compare the efficacy of low dose catheter directed thrombolysis (CDT) to unfractioned heparin (UFH) in patients with intermediary-high risk pulmonary embolism (PE).

Patients (n=60) with acute intermediary-high risk PE will be randomized 1:1 to UFH (bolus 80 international units per kilo (IU/kg)) followed by 18 IU/kg/hour until activated partial thromboplastin time (APTT) is 2-2.5 of reference value) or CDT (4mg alteplase (r-tPA) per catheter, infusion over 2 hours) in an open label, outcome assessor blinded, randomized, controlled trial. Primary efficacy endpoint is improvement in right-/left ventricular ratio 24 hours after randomization. Secondary endpoints are 30 days mortality, recurrent PE, length of hospital stay and reduction in thrombus burden evaluated by pulmonary CT angio. Safety endpoints are minor and major bleedings.

DETAILED DESCRIPTION:
1. Aim To investigate if low dose catheter directed fibrinolysis for 2 hours is superior to unfractioned heparin with regards to unloading the right ventricle in acute intermediate-high risk pulmonary embolism
2. Methods 2.1 Study design The study is an open label, randomized, single center trial. Patients (n=60) with acute intermediate-high risk acute pulmonary embolism diagnosed with computed tomography pulmonary angiography (CTA) will be treated with unfractionated heparin (UFH) at the time of diagnosis and randomized 1:1 within 48 h to low dose catheter directed thrombolysis or continuation of UFH. Primary endpoint is improvement in right-to-left ventricular ratio (RV/LV ratio) evaluated by CTA 24 hours (±2h) after randomization. Secondary endpoints are 30 day mortality, reduction in thrombus burden evaluated by CTA, length of hospital stay and recurrent PE. Safety will be monitored as minor and major bleeding.

   2.2 Patients Patients are eligible for inclusion if they apply to all inclusion and none of the exclusion criteria and give their informed written consent

   2.2.1 Recruitment and informed consent Patients admitted to a hospital in Region Midt with acute pulmonary embolism will be screened for eligibility for inclusion in the trial by a local investigator at the day of admission. The local investigator will then contact the PI that will ensure that the patient is eligible for inclusion. All patients referred for possible inclusion will be registered as screened. If eligible for inclusion, the local investigator will give the verbal and written study information to the patient. The local investigator will do the best possible to avoid interruptions and the staff will be informed accordingly to ensure fewest possible interruptions during the verbal information. The patient will be informed that it is possible to have an assessor during the verbal information. After verbal and written information the patient will be given a minimum of 1/2 hour and up to 8 hours for reflection before giving their consent. The patient will also be informed, that they can withdraw their consent at any time.

   2.2.2 Benefits, risk and safety The patients included in this trial will be treated with the highest known standard of care for their acute PE. If randomized to conventional treatment (UFH), there is no obvious benefit for the individual patient with regards to treatment, but the extra diagnostics may aid the treating physician to optimize their standard treatment. For patients randomized to CDT there is a potential benefit of treatment due to faster removal of thrombus mass in the pulmonary arteries. The biggest advantage of this trial is for future patients with acute PE, as this trial will aid future decisions with regards to treatment with CDT or UFH. Safety is discussed in section 12.

   2.2.3 Patient discontinuation and substitution Patients that are included in the study but discontinue (any cause) before their follow-up CTA 24 hours after treatment will be excluded from the final data analysis and substituted by a new study patient. Data from patients that discontinue (any cause) after their follow-up 24 hours CTA will be included in the final analysis. Data from patients that withdraw their consent for study participation will be excluded and substituted by a new study patient, if the trial is still ongoing at time of withdrawal.

   2.3 Treatment and Randomization 2.3.1 Randomization After study inclusion, patients will be transferred to Department of Cardiology, Aarhus University Hospital. Then, patients will be randomized to continue UFH with or without CDT. Patient data will be registered in the online case report form (CRF) hosted in a RedCap database and the RedCap database tool for randomization will be used for randomization to treatment. The recorded variable are listed in appendix 1.

   2.6 Statistics A previous similar study using ultrasound assisted CDT (10-20 mg rt-PA over 15 hours) versus UFH ULTIMA found an improvement in RV/LV ratio of -0.3 (SD, 0.2) vs. -0.03 (SD, 0.16) with UFH alone. And the OPTALYSE(6) study found an improvement in RV/LV ratio of -0.46 (no SD reported, only abstract published) using 4/8 mg rt-PA over 2 hours. Using the most conservative result from the previous trials with a RV/LV difference of 0.17 between groups, and SD from a current unpublished PE study from our institution of 0.3, power of 0.8 and a significance level of 0.05 the sample size is calculated to be 21 patients in each treatment group. Based on this power calculation we plan to include a total of 60 patients randomized 1:1 with an interim analysis after the inclusion of 42 patients. All data with dichotomous outcome will be analyzed using the fisher's exact test. Between group comparison of continuous data will be compared using the two-sided unpaired t-test or Wilcoxon rank sum test. Within group comparison of continues data will be performed using the two-sided paired t-test and ordinal data with the Wilcoxon signed-rank test. Ordinal data between groups will be analyzed using a chi-square test. Data will be analyzed as intention to treat.
3. Time Schedule In Region Midt, 350 patients with PE is admitted to the hospital each year. Based on a previous study at our institution including patients with intermediary-high risk PE patients we plan to include 20 patients/year over a 3 year period.
4. Feasibility The Dep. of Cardiology, Aarhus University Hospital have a long tradition of including patients in randomized trials. All necessary equipment and personnel for the study is available at the department. Associate Professor Asger Andersen, MD, PhD (AA) and Professor Jens Erik Nielsen-Kudsk, MD, DMSc (JENK) will be principal investigators.
5. Ethics The study will adhere to Danish laws of ethics and management of personal data. The study will not begin before it have been approved by The regional data monitoring board, the Regional Ethics Committee and the Danish Medicines Agency. The study will adhere to the standards of good clinical practice and it will be monitored by the Unit of "Good Clinical Practice" at Aalborg and Aarhus University Hospitals. The study will pay the outmost respect to the included patients mental and physical health and their personal integrity.
6. Safety The treatment is considered safe and previous studies suggest that this approach may be better than conventional therapy. All patients will be monitored continuously with ECG, blood pressure and clinical status in the catheterization laboratorium and after return to the ward with blood pressure, pulse, respiratory frequency and clinical status minimum every hour until two hours after termination of alteplase infusion. If any suspected or confirmed complication occurs the physician on call, attending the ward, will be contacted to initiate relevant diagnostic testing and/or treatment. The staff and physicians attending the ward are well trained in attending critically ill patient including patients with acute PE and patients that have been catheterized. The invasive procedure will be performed by a trained invasive cardiologist whose expertise is to catheterize the pulmonary circulation. Using the low dose short period regime suggested in this protocol there have not been reported any bleedings in clinical studies. The patients included in the trial will be exposed to an extra CTA which exposes the patient to 4-8 millisievert which approximates the background radiation a person receives over 3 years and increases the risk of a fatal cancer from 25% to 25.045%. Patients randomized to CDT will receive an additional 1-2 millisievert from the fluoroscopy. The patients included in this study have an estimated 30 day mortality of 15% and solid preliminary data suggest the treatment to be effective and safe. Therefore it is the investigators opinion that the benefits of doing this study outweighs the risks.
7. Publication The results from this trial will be published whether negative, neutral or positive. First author will be AA and last author JENK. Members of the steering committee and responsible investigators from each trial site will be co-authors. Other contributing members of the trial will be offered co-authorship if their contribution adheres to the Vancouver protocol for co-authorship.
8. Perspectives This study will be the first randomized trial to investigate if low dose catheter based thrombolysis is superior to unfractioned heparin with regards to unloading the right ventricle in patients with acute intermediate-high risk pulmonary embolism. If efficient, the findings from this study may motivate a larger clinical trial with hard clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 and < 81 years
* Debut of symptoms <14 days
* Acute symptomatic Intermediate-high risk pulmonary embolism (PE, according to 2014 European Society of Cardiology guidelines) confirmed by computed tomography angiography (CTA) with the embolus located in at least one proximal lower lobe or main pulmonary artery.
* Right-to-left ventricular dimension ratio >1.0 on CTA or trans-thoracic echocardiography (TTE)

Exclusion Criteria:

* Significant bleeding risk or other contraindications to catheter directed thrombolysis (CDT) or unfractionated heparin*
* Not possible to perform CDT within 48 hours after diagnosis
* Pregnancy
* Cardiac arrest requiring cardiopulmonary resuscitation
* Life expectancy < 120 days
* Altered mental status such that the patient is unable to provide informed consent
* Suspected or known chronic thromboembolic pulmonary hypertension
* Sustained hypertension (>180 mmHg systolic and/or >105 mmHg diastolic)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Right ventricle divided by left ventricular diameter (RV/LV ratio) | 24 hours after intervention
  Measured on ECG gated contrast enhanced computed tomography

SECONDARY OUTCOMES:
Reduction in thrombus burden | 24 hours after intervention
  A modified miller index till be measured on ECG gated contrast enhanced computed tomography
Thirty day mortality | 30 days after intervention
  The number of patients that are decease within 30 days after the intervention will be assessed from the patient files.
Length of hospital stay | 3 months after intervention
  The length of hospital stay in days will be evaluated from the patient files
Recurrent pulmonary embolism | 3 months after intervention
  Number of patients with recurrent pulmonary embolism will be evaluated from the patient files
Lung perfusion | 24 hours after intervention
  Lung perfusion will be evaluated and quantified with dual energy computed tomography

OTHER OUTCOMES:
Minor and major bleeding | 24 hours after intervention
  Bleeding events will be recorded during the hospital stay during the daily rounds

CONTACTS AND LOCATIONS:
Overall Officials: Asger Andersen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Dep. Cardiology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Sogaard KK, Schmidt M, Pedersen L, Horvath-Puho E, Sorensen HT. 30-year mortality after venous thromboembolism: a population-based cohort study. Circulation. 2014 Sep 2;130(10):829-36. doi: 10.1161/CIRCULATIONAHA.114.009107. Epub 2014 Jun 26. PMID 24970783
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Engelberger RP, Spirk D, Willenberg T, Alatri A, Do DD, Baumgartner I, Kucher N. Ultrasound-assisted versus conventional catheter-directed thrombolysis for acute iliofemoral deep vein thrombosis. Circ Cardiovasc Interv. 2015 Jan;8(1):e002027. doi: 10.1161/CIRCINTERVENTIONS.114.002027. PMID 25593121